CLINICAL TRIAL: NCT00138814
Title: A Randomised Comparison of Breast Conservation With or Without Lumpectomy Radiotherapy Boost
Brief Title: Boost Use in Breast Conservation Radiotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St George Hospital, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 96/84 Graham
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2005-12-15 (Estimated); Status verified 2005-09

CONDITIONS: Breast Neoplasms
Keywords: Neoplasm recurrence, local; Radiotherapy dosage; Cosmesis; Mastectomy, segmental
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Recurrence, Local | interventions — Radiotherapy

INTERVENTIONS:
Procedure: Radiotherapy (boost versus no boost)

SUMMARY:
This is a two arm randomized study for patients who are undergoing radiotherapy following breast conservation surgery for breast cancer. Local recurrence of breast cancer will be compared for patients receiving boost or no boost radiotherapy.

DETAILED DESCRIPTION:
A boost dose of radiation is commonly but not universally employed in breast conservation techniques.

The potential disadvantages when a boost is employed include:

* Increased complexity of treatment
* Increased duration of treatment
* Increased travel, social/employment dislocation
* Increased complications
* Worse cosmesis and/or increased breast discomfort
* Increased difficulty in detecting recurrence.
* Prolongation of gap or increased delay for chemotherapy if indicated

The potential advantages of a boost are the following:

* Reduced local failure rates
* Reduced local failure translating to improved survival
* Maximising cosmesis by reducing dose to larger breast volume

None of the potential advantages have been clearly demonstrated in a controlled fashion although there are sound theoretical reasons that a boost will improve local control. Holland's landmark paper using radiologic-pathologic correlation of mastectomy specimens, whilst finding residual foci beyond the boundaries of cosmetically acceptable resection margins, also found most of the residual tumour relatively close to the index mass. There is a known dose-response for control of breast cancer. Kurtz reported a doubling of the longterm recurrence rate when the dose to the tumour bed was less than 75 Gy or delivered at less than 8 Gy per week from 15% to 30% using telecesium following lumpectomy. Treating the entire breast to doses above 50 to 54 Gy in 5 weeks is associated with significantly worse cosmesis, hence the common use of a boost. There are as yet no controlled comparisons published however Beadle reported a 50% increase in the rates of poor cosmesis when a boost was employed. Borger has demonstrated that the risk of fibrosis increases fourfold with every 100 cm3 increase in boost volume. Accurate localisation of the tumour bed for boost delivery is difficult in the absence of radioopaque clips (uncommonly employed by our referral base). The use of electrons to deliver the boost has been reported to decrease the cosmetic outcome compared to I192 because of telangiectasia, although this is controversial with other reports indicating superior results with electrons, which is the modality available at St George and Wollongong. The latter avoids hospitalisation. There is at least one other randomised multicentre study being conducted testing the value of a boost by the EORTC in Europe but no results are yet available.

Comparisons: Patients will be stratified by chemotherapy (none, AC, non-AC) and within the non-AC arm will be randomised in respect to timing (pre, sandwich, concurrent) of radiotherapy. Randomisation to treatment will be - boost (45Gy 25# + 16Gy 8#) or no boost (50Gy 25#).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven carcinoma of the breast, T1-2 (0-5cm) N0-1, M0.
* Pure ductal carcinoma in situ accepted if completely excised.
* Any receptor status.
* Extensive intraductal cancer (EIC) accepted if completely excised.

Exclusion Criteria:

* Unable to consent
* Vascular/collagen disorder
* Prior malignancy except minor skin squamous cell or basal cell carcinoma or carcinoma in-situ of the cervix .
* Gross multifocal disease
* Involvement of margins.
* Bilateral breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680
Dates: Start 1997-01; Study Completion 2015-12

PRIMARY OUTCOMES:
Local failure of breast cancer at 72 month median follow-up and 10 year median follow-up for final analysis

SECONDARY OUTCOMES:
Local control translating to survival over 10 year median follow-up
Quality of life at yearly intervals with reference to baseline
Breast cosmesis - patient assessment and photos

CONTACTS AND LOCATIONS:
Overall Officials: Associate Prof. Peter H Graham, MBBS FRANZCR, Principal Investigator — Cancer Care Centre, St George Hospital, Sydney, Australia; Dr Geoff Delaney, MBBS FRANZCR, Principal Investigator — Liverpool Hospital, Sydney, Australia; Dr Chris Fox, MBBS FRANZCR, Principal Investigator — Wollongong Hospital, Wollongong, Australia
Locations (3):
- Australia (3):
  - Liverpool Hospital, Sydney, New South Wales
  - Cancer Care Centre, St George Hospital, Sydney, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales

REFERENCES:
- [Derived] Browne LH, Graham PH. Good intentions and ICH-GCP: Trial conduct training needs to go beyond the ICH-GCP document and include the intention-to-treat principle. Clin Trials. 2014 Dec;11(6):629-34. doi: 10.1177/1740774514542620. Epub 2014 Jul 14. PMID 25023199
- [Derived] Hau E, Browne L, Capp A, Delaney GP, Fox C, Kearsley JH, Millar E, Nasser EH, Papadatos G, Graham PH. The impact of breast cosmetic and functional outcomes on quality of life: long-term results from the St. George and Wollongong randomized breast boost trial. Breast Cancer Res Treat. 2013 May;139(1):115-23. doi: 10.1007/s10549-013-2508-z. Epub 2013 Apr 12. PMID 23580069
- [Derived] Hau E, Browne LH, Khanna S, Cail S, Cert G, Chin Y, Clark C, Inder S, Szwajcer A, Graham PH. Radiotherapy breast boost with reduced whole-breast dose is associated with improved cosmesis: the results of a comprehensive assessment from the St. George and Wollongong randomized breast boost trial. Int J Radiat Oncol Biol Phys. 2012 Feb 1;82(2):682-9. doi: 10.1016/j.ijrobp.2010.11.025. Epub 2011 Jan 20. PMID 21255943
- [Derived] Millar EK, Graham PH, O'Toole SA, McNeil CM, Browne L, Morey AL, Eggleton S, Beretov J, Theocharous C, Capp A, Nasser E, Kearsley JH, Delaney G, Papadatos G, Fox C, Sutherland RL. Prediction of local recurrence, distant metastases, and death after breast-conserving therapy in early-stage invasive breast cancer using a five-biomarker panel. J Clin Oncol. 2009 Oct 1;27(28):4701-8. doi: 10.1200/JCO.2008.21.7075. Epub 2009 Aug 31. PMID 19720911